CLINICAL TRIAL: NCT06141876
Title: A Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability and Efficacy of Psilocybin-Assisted Psychotherapy in Treating Severe Depression Among Adults With Post-Traumatic Stress Disorder (PTSD).
Brief Title: Evaluation of Psilocybin-Assisted Psychotherapy in Treating Severe Depression in Patients With PTSD
Acronym: SUMMIT-90
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Apex Labs Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: APEX-002-A02-01
Record Dates: First submitted 2023-11-08; First posted 2023-11-21 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Post-traumatic Stress Disorder; Depression
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression | interventions — Psilocybin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): APEX-002-A02
  Interventions: Drug: APEX-002-A02
- Placebo (Placebo Comparator): matched placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: APEX-002-A02 — Active
  Other Names: psilocybin
  Arms: Active
Other: Placebo — placebo
  Arms: Placebo

SUMMARY:
Post-Traumatic Stress Disorder (PTSD) is a mental disorder that may develop in people who have been exposed to a traumatic event, including actual or threatened death, serious injury, or sexual violence. Exposure to a traumatic event is defined as directly experiencing the event, learning about the event, or repeated exposure to details of the event. PTSD is often accompanied by other psychiatric and physical comorbidities, both of which are associated with elevated healthcare costs. Depression, psychosis and suicide rates are consistently reported in greater proportion of PTSD patients. Despite the overwhelming impact of PTSD and comorbid depression, there is a shortfall of effective treatments with few side effects that target the broad range of symptoms, including depression.

Psilocybin has been studied for the treatment of depression, anxiety, tobacco and alcohol use disorders, obsessive-compulsive disorder, end of life depression and anxiety, demonstrating safety and efficacy for a variety of indications, with no significant adverse events occurring during the course of treatment and follow-up. Notably, in a participant group distinguished by long-standing, moderate to severe major depressive disorder, two doses of psilocybin-assisted therapy were found to be as effective in antidepressant effects as 6 weeks of daily escitalopram, a commonly used SSRI. Promising results found in these studies have led to psilocybin recently receiving breakthrough designation from the US FDA for its potential therapeutic effect in the treatment of depression.

Based on previous research, psilocybin has demonstrated a favorable safety profile and has shown preliminary efficacy against depression as well as other symptoms that typically affect patients with PTSD. Unlike traditional SSRIs which are associated with treatment-resistance and addiction, psilocybin requires few doses to improve a wide-range of symptoms and has not been linked with physical dependence. Furthermore, the effect of other psychedelics can vary greatly and may potentially exacerbate existing conditions.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals between 18 and 65 years of age, inclusive, at the time of consent.
2. Individuals who are fluent in the language of the study site, specifically English or French.
3. Meet DSM-5 criteria for current PTSD with presence of symptoms for at least 6 months at screening.
4. Participant must have at least moderate PTSD, as scored as ≥35 on the CAPS-5 scale at screening.
5. Participant must have severe depression, as scored as ≥30 on the BDI-II scale at screening.
6. If individuals are on psychotropic medications, they must be on stable doses (no dosing adjustments/changes for ≥4 weeks) prior to beginning of the study and for the duration of the study.
7. If individuals are users of psychoactive substances, including alcoholic beverages, tobacco, and cannabis, they must remain on stable doses for the duration of the study.
8. For individuals of childbearing potential involved in any sexual intercourse that could lead to pregnancy: willing to use adequate birth control to prevent pregnancy (in participant or partner) for the entire duration of the study.
9. Capable of providing ongoing, signed informed consent.
10. Available for the duration of the study, and able and willing to comply with all study procedures, including completion of questionnaires.
11. Agree to identify a local contact person to the research team, that is available over the entire course of the subject's participation in the study to act as an emergency contact.

Exclusion Criteria:

1. Female subject that is pregnant, is planning or suspected to become pregnant, or is lactating.
2. Known or suspected hypersensitivity or contraindication to psilocybin or any constituents or excipients of the study drug.
3. Abnormal and clinically significant results on the physical examination, vital signs, ECG or laboratory tests at screening.
4. Presence of any unstable medical condition or neurological illness, in the opinion of the Investigator.
5. History of clinically significant cardiovascular disease including but not limited to stroke, myocardial infarction or clinically significant arrhythmia (in the past 1 year).
6. Indication of inadequately treated current hypertension (resting systolic blood pressure >140 mmHg and/or diastolic blood pressure >90 mmHg) at screening.
7. If a subject is being treated with inhibitor(s) of UGT1A9, UGT1A10, monoamine oxidase (MAO), aldehyde dehydrogenase (ALDH), or alcohol dehydrogenase (ADH) they should be discontinued at least five half lives prior to administration of study drug.
8. Lifetime history of psychosis-related disorder or bipolar disorder (I or II).
9. Subject has 1st degree relative(s) with schizophrenia or bipolar disorder.
10. At the time of screening, any condition other than PTSD judged to be the primary presenting psychiatric diagnosis, in the opinion of the Investigator.
11. Clinical diagnosis of dementia or any physical, cognitive, or language impairment of such severity as to adversely affect the validity of the data derived from the patient reported outcomes.
12. History of any other clinically significant pulmonary, gastrointestinal, hepatic, renal or any other major concurrent illness that, in the opinion of the investigator, may interfere with the interpretation of the study results or constitute a health risk for the participant if he/she takes part in the study.
13. Individuals who present a current risk to themselves or others, as assessed by the Investigator. This includes, but is not limited to:

    1. Active suicidal ideation with specific plan and intent in the past 1 month, as assessed with the C-SSRS at screening.
    2. History of suicidal behavior (actual attempt, interrupted attempt, aborted or self-interrupted attempt, preparatory acts or behavior) in the past 3 months, as assessed with the C-SSRS at screening.
    3. Any prior suicidal ideation/behavior that, per the Investigator's judgment, makes the participant unsuitable for the study.
14. Current active Substance Use Disorder or Alcohol Use Disorder, as assessed by the Investigator via medical screening.
15. Individuals with other personal circumstances and behaviour judged to impact safety (risk and not be able to adhere to the protocol requirements).
16. Individuals with significant prior exposure to psilocybin, defined as:

    1. Chronic use (>10 exposures) of psilocybin in any form and at any dose in the past year; OR
    2. Any use of psilocybin within 4 weeks prior to screening; OR
    3. Any previous use of psilocybin for PTSD or related symptoms, including depression, that was discontinued due to lack of effect, as judged by the individual or their treating physician.
17. Self reported use within 12 weeks prior to screening of (i) classical psychedelics other than psilocybin (LSD, mescaline, dimethyltryptamine); (ii) MDMA; (iii) ketamine, and; (iv) dextromethorphan.
18. Actively participating in other interventional clinical trial(s).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2023-12-15 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-06-15 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Baseline to Day 140
  Treatment emergent AEs and SAEs
Number of participants with abnormal vital signs, abnormal physical exam findings, abnormal ECG, and abnormal laboratory tests results | Baseline to Day 140
  Measurements: vital signs, physical exam, ECG, and laboratory tests
Change in severity of depressive symptoms | Baseline to Day 77
  Assessed by total score of Beck Depression Inventory (BDI-II); 21-items scale. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.

SECONDARY OUTCOMES:
Change in severity of depressive symptoms | Baseline to Days 21, 49, and 140
  Assessed by total score of Beck Depression Inventory (BDI-II); 21-items scale. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
Change in severity of PTSD symptoms | Baseline to Days 21, 49, 77 and 140
  Assessed by total score of Clinician-Administered PTSD Scale for Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (CAPS-5); 30-item questionnaire. Severity rating: 0=absent, 1-mild/sub-threshold, 2-moderate/threshold, 3-severe/markedly elevated, 4-extreme/incapacitating.
Change in severity of anxiety | Baseline to Days 21, 49, 77 and 140
  Assessed by Beck Anxiety Inventory (BAI); 21-item scale. BAI scores are classified as minimal anxiety (0 to 7), mild anxiety (8 to 15), moderate anxiety (16 to 25), and severe anxiety (30 to 63).
Change in presence and severity of suicidal ideation and behaviour | Baseline to Days 21, 49, 77 and 140
  Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS); 10-category scale with binary (yes/no) responses. There are no specified clinical cutoffs for the C-SSRS due to the binary nature of the responses to items. When an item is endorsed ("yes"), the clinician must pose follow-up inquiries to obtain additional information.
Change in chronic pain severity | Baseline to Days 21, 49, 77 and 140
  Assessed by Brief Pain Inventory (BPI); 9-point questionnaire with 0-10 scale for each point; 0=no pain, 10=pain as bad as you can imagine.

IPD SHARING:
Plan to Share IPD: Undecided